CLINICAL TRIAL: NCT00993213
Title: Mechanisms Defending Fat Mass in Humans After Lipectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical Nutrition Research Unit-Metabolic and Energy Balance Laboratories (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-499; R01DK061668 (NIH)
Record Dates: First submitted 2009-10-08; First posted 2009-10-12 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Disproportionate Shape; Expanded Fat Pads
Keywords: fat mass; body composition
MeSH Terms: interventions — Standard of Care; Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposuction (Active Comparator): Standard of Care with Liposuction
  Interventions: Procedure: Standard of Care with Liposuction
- No Liposuction (Sham Comparator): Standard of Care without Liposuction'
  Interventions: Other: Standard of Care without Liposuction

INTERVENTIONS:
Procedure: Standard of Care with Liposuction — Standard of Care encompasses body composition measurements, a euglycemic clamp and fat biopsies, followed by Liposuction surgery.
  Arms: Liposuction
Other: Standard of Care without Liposuction — Standard of Care encompasses body composition measurements, a euglycemic clamp and fat biopsies. Liposuction surgery will not be performed.
  Arms: No Liposuction

SUMMARY:
Liposuction surgery is common, yet animal and limited human data suggest that fat returns when removed. This study was designed as a 1-year randomized-controlled trial of suction lipectomy versus no intervention to determine if adipose tissue is defended, and if so to determine the anatomic pattern of redistribution.

DETAILED DESCRIPTION:
Specific Aims:

1. To determine if suction lipectomy fails to modify regional and/or total body fat over three years.
2. To determine if the expression of candidate genes predicts and/or relates to subcutaneous adipose tissue growth or depletion in subcutaneous adipose tissue after suction lipectomy.
3. To examine adipose tissue before and after suction lipectomy to uncover novel genes where expression predicts and/or relates to subcutaneous adipose tissue growth or depletion after subcutaneous suction lipectomy.

ELIGIBILITY:
Inclusion Criteria:

* Eligible premenopausal women between the ages of 18-50 years;
* BMI of 22-27 kg/m2 at the subjects maximum body weight;
* Weight stable for at least 3 months (defined as a <5-7% change from the maximum weight over 3-6 months);
* Non-smokers.

Exclusion Criteria:

* Any history of glucose intolerance, dyslipidemia, liver, kidney and cardiac disease, hypertension, cancer or any other chronic debilitating disorder that might have interfered with a 'normal' lifestyle, e.g. nutrition, physical activity;
* Thyroid hormone replacement with abnormal thyroid stimulating hormone (TSH) results;
* Use of oral contraceptives if the subject did/could not remain on therapy throughout study participation.
* Reduced-obese, defined as a history of:

  1. obesity and weight loss >10% of maximum body weight, or
  2. liposuction or gastric bypass surgery;
* Evidence of body dysmorphic disorder;
* Taking sex steroids, glucocorticoids, or medications affecting carbohydrate and lipid metabolism;
* Hematocrit, hemoglobin, white blood cell count (WBC), platelet count, liver or renal function tests out of the normal range;
* Fasting plasma glucose >110 mg/dL;
* Triglycerides >200 mg/dL;
* High density lipoprotein (HDL) cholesterol <35 mg/dL;
* Low density lipoprotein (LDL) cholesterol >160 mg/dL;
* Proteinuria;
* Blood pressure >140/90 mm/Hg;
* Electrocardiogram abnormalities;
* History of claustrophobia;
* Placement of metal implants*
* History of internal metal fragments*

*Were evaluated by the radiologist prior to study determination*

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2004-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Changes in body composition. | Baseline, 6wks, 6mos, 1-year
  Changes in body composition as measured by Dual X-ray Absorptiometry (DXA).

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Eckel, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Background] Wu X, Zvonic S, Floyd ZE, Kilroy G, Goh BC, Hernandez TL, Eckel RH, Mynatt RL, Gimble JM. Induction of circadian gene expression in human subcutaneous adipose-derived stem cells. Obesity (Silver Spring). 2007 Nov;15(11):2560-70. doi: 10.1038/oby.2007.308. PMID 18070747
- [Result] Hernandez TL, Kittelson JM, Law CK, Ketch LL, Stob NR, Lindstrom RC, Scherzinger A, Stamm ER, Eckel RH. Fat redistribution following suction lipectomy: defense of body fat and patterns of restoration. Obesity (Silver Spring). 2011 Jul;19(7):1388-95. doi: 10.1038/oby.2011.64. Epub 2011 Apr 7. PMID 21475140